CLINICAL TRIAL: NCT06932146
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamic (PD) Effects of LLX-424 in Patients With a History of Kidney Stones
Brief Title: A Phase 2a Study of LLX-424 in Patients With a History of Kidney Stones
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lilac Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LLX-002
Record Dates: First submitted 2025-04-02; First posted 2025-04-17 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Kidney Stones
Keywords: oxalate; glycolate oxidase
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LLX-424 (Experimental): Tablets for oral administration
  Interventions: Drug: LLX-424
- Placebo (Placebo Comparator): Tablets for oral administration
  Interventions: Drug: LLX-424

INTERVENTIONS:
Drug: LLX-424 — Tablets for oral administration
  Other Names: glycolate oxidase inhibitor

SUMMARY:
This is a Phase 2a study of glycolate oxidase inhibitor LLX-424 in patients with a history of kidney stones. Eligible subjects with a history of kidney stones will be randomized to receive study drug (LLX-424 or placebo) for 8 weeks.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled study designed to assess the safety, tolerability, PK, and PD effects of LLX-424 in patients with a history of kidney stones.

Following completion of screening procedures, on Study Day 1, eligible subjects will be randomized in a 2:1 ratio to receive either LLX-424 or matching placebo, respectively.

An outpatient safety Follow-up Visit will be scheduled on Day 63 or 7 days after the last dose (end of study visit).

ELIGIBILITY:
Inclusion Criteria:

* History of kidney stones documented in medical records
* 24-hour urine oxalate excretion
* Body mass index 18.5 to 38 kg/m2 inclusive
* Estimated glomerular filtration rate ≥ 60 mL/min/1.73m2

Exclusion Criteria:

* History or medical record evidence of kidney stones that are not calcium oxalate
* Unstable kidney function
* Spot urine protein to creatinine ratio ≥ 1 mg/mg at screening
* History of kidney transplantation
* Hemoglobin A1c > 9.5% at screening
* History of enteric hyperoxaluria, intestinal malabsorption, bariatric surgery, intestinal surgery, inflammatory bowel disease
* History or evidence of cirrhosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2025-03-23 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | From the first dose and for up to 9 weeks
  Percentage of subjects with TEAEs
Percentage of subjects with study drug-related severe laboratory-based AEs | From the first dose and for up to 9 weeks
  Laboratory-based adverse events
QT interval on ECG | From the first dose and for up to 9 weeks
  Percentage of subjects with an increase from baseline in the QTcF by > 60 milliseconds

SECONDARY OUTCOMES:
Mean change from baseline in 24-hour urine oxalate excretion rate | From pre-dose to Study Day 56
  Comparison between LLX-424 group and the placebo group
Peak plasma concentration (Cmax) of LLX-424 | From pre-dose to Study Day 56
  Cmax of plasma LLX-424
Area under the curve (AUC) of plasma LLX-424 concentration versus time after dosage | From pre-dose to Study Day 56
  AUC of plasma LLX-424
Peak plasma concentration (Cmax) of glycolate | From pre-dose to Study Day 56
  Cmax of plasma glycolate
Area under the curve (AUC) of plasma glycolate concentration versus time after dosage | From pre-dose to Study Day 56
  AUC of plasma glycolate

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Research Site #2, Saint Paul, Minnesota
  - Clinical Research Site #3, Springfield, Missouri
  - Clinical Research Site #1, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://www.lilactx.com